CLINICAL TRIAL: NCT00751062
Title: A 6-month, Randomized, Double-masked Comparison of PhXA41 With Timolol in Patients With Open Angle Glaucoma or Ocular Hypertension. A Multi-centre Study in Scandinavia
Brief Title: A Study of Open Angle Glaucoma or Ocular Hypertension in Patients Within Scandinavia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9200PG006; A6111130
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-09

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: open angle glaucoma ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Timolol; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timolol (Active Comparator)
  Interventions: Drug: timolol
- PhXA41 (Experimental)
  Interventions: Drug: PhXA41

INTERVENTIONS:
Drug: timolol — One drop in the affected eye every morning from the morning bottle and one drop every evening from the evening bottle.
  Arms: Timolol
Drug: PhXA41 — One drop in the affected eye every morning from the morning bottle and one drop every evening from the evening bottle
  Arms: PhXA41

SUMMARY:
PhXA41 is not inferior to timolol in reducing intra-ocular pressure

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral primary open angle glaucoma, capsular glaucoma, pigmentary glaucoma or ocular hypertension.
* Open angle glaucoma appearing more than 6 months after cataract surgery is recognized as primary open angle glaucoma. (individuals requiring treatment bilaterally must fulfill eligibility criteria for both eyes.)
* IOP of 22mmHg or higher obtained during the pre-study period.

Exclusion Criteria:

* History of acute angle closure.
* Severe trauma at any time.
* Intraocular surgery or argon laser trabeculoplasty within 6 months.
* Current use of contact lenses.
* History of severe dry eye syndrome.
* Ocular inflammation/infection with three months of inclusion.
* Any condition preventing reliable applanation tonometry.
* Unacceptable finding at pre-study ocular examination as specified in the Case Report Forms.
* In Investigator regards monotherapy insufficient with respect to optic nerve head and/or visual field status.
* Treatment of elevated IOP with any topical B-adrenergic antagonist regularly for a period longer than 3 months and/or treatment at any time during 6 months prior to study start.
* Cardiac failure, sinus bradycardia, second and third degree of atrio-ventricular block.
* Bronchial asthma, history of bronchial asthma or chronic obstructive pulmonary disease.
* Having participated in any other clinical study within the last month.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 1992-11; Primary Completion 1993-12 (Actual); Study Completion 1993-12 (Actual)

PRIMARY OUTCOMES:
to demonstrate the IOP-reducing effect of PhXA41 is comparable to that of timolol at the end of 6 months of treatment. | 6 mos

SECONDARY OUTCOMES:
to demonstrate the IOP-reducing effect of PhXA41 administered in the morning is equivalent the effect of PhXA41 administered in the evening | 6 mos

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Denmark (2):
  - Pfizer Investigational Site, Hellerup
  - Pfizer Investigational Site, Vejle
- Pfizer Investigational Site, Oulu, Finland
- Norway (3):
  - Pfizer Investigational Site, Bergen
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Trondheim
- Sweden (7):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Huddinge
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Umeå
  - Pfizer Investigational Site, Uppsala

REFERENCES:
- [Derived] Varma R, Hwang LJ, Grunden JW, Bean GW, Sultan MB. Assessing the efficacy of latanoprost vs timolol using an alternate efficacy parameter: the intervisit intraocular pressure range. Am J Ophthalmol. 2009 Aug;148(2):221-6. doi: 10.1016/j.ajo.2009.02.035. Epub 2009 May 9. PMID 19427617
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=9200PG006&StudyName=A%20study%20of%20open%20angle%20glaucoma%20or%20ocular%20hypertension%20in%20patients%20within%20Scandinavia